CLINICAL TRIAL: NCT05648474
Title: Advanced Techniques in Intraoperative Monitoring for the Lateral Lumbar Interbody Fusion Procedure: a Utility Study
Brief Title: Intraoperative Monitoring for the Lateral Lumbar Interbody Fusion Procedure
Status: Recruiting | Type: Observational
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ATEC.AI-2001
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Intervertebral Disc Degeneration; Stenosis, Spinal; Spondylolisthesis; Spinal Deformity; Spinal Instability
Keywords: Spine; Surgery; Adult; Neuromonitoring; Electromyography; Somatosensory evoked potentials
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis | interventions — Evoked Potentials, Somatosensory; Monitoring, Intraoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult undergoing 1- or 2-level lateral lumbar interbody fusion surgery, inclusive of the L4-5 level
  Interventions: Diagnostic Test: Somatosensory evoked potential [SSEP] intraoperative monitoring

INTERVENTIONS:
Diagnostic Test: Somatosensory evoked potential [SSEP] intraoperative monitoring — No study specific intervention is performed. Intraoperative neuromonitoring system that is observed in this study is for assessing the health of the lumbar plexus during lateral lumbar interbody fusion surgery

SUMMARY:
This study is designed to evaluate the clinical utility of a known intraoperative neuromonitoring modality (SSEP) using saphenous nerve as the site of stimulation to identify changes to the lumbar nerves which may be at risk during the lateral lumbar interbody fusion (LLIF) procedure.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of planned surgery.
* Indicated for 1- or 2-level instrumented LLIF surgery (in either prone or lateral decubitus positions), inclusive of the L4-5 disc space.
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Patients requiring surgical treatment at more than 2 lumbar levels.
* Patients with peripheral neuropathy such as from diabetes or other conditions that might affect the reliability of intraoperative neuromonitoring.
* Patients with prior history of partial/full hip or knee joint replacement surgery (i.e., arthroplasty or resurfacing) on the leg targeted for saphenous monitoring and electrode placement.
* Patients with presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Female patients who are pregnant or wanting to become pregnant during the timeframe of study participation.
* Patients participating in another clinical study which may compromise this study's results or compliance with this study's procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes undergoing LLIF surgery atone or two levels inclusive of the L4-5 level.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of SSEP neuromonitoring in post-operative clinical diagnosis of motor/sensory deficits | 6 weeks or until new or worsened neural deficits are resolved, but not exceeding 12 months.
  This outcome measure determines the utility of the saphenous nerve SSEP monitoring based on the correlation of intraoperative neuromonitoring results with new or worsened postoperative neural deficits, as measured by motor and sensory physical exam.

SECONDARY OUTCOMES:
Determination of the positive predictive value (PPV) and negative predictive value (NPV) of free run and SSEP monitoring modalities. | 6 weeks or until new or worsened neural deficits are resolved, but not exceeding 12 months.
  This outcome measure includes:
  * Correlating specific monitoring findings with incidence of new or worsened motor or sensory deficits post-operatively and their correlation with patient-specific and surgical factors.
  * Correlating patient and surgical factors with new and worsened postoperative neural deficits.

CONTACTS AND LOCATIONS:
Locations (1):
- Alphatec Spine Inc., Carlsbad, California, United States